CLINICAL TRIAL: NCT04982094
Title: Counting On U: Supporting SME Advisors and Owners Towards Better Mental Health
Brief Title: Counting On U: Towards Better Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leanne Saxon (Other)
Collaborators: Institute of Public Accountants (Unknown); Beyond Blue (Unknown); WorkSafe Victoria (Unknown); Mental Health First Aid Australia (Unknown)
Responsible Party: Sponsor-Investigator, Leanne Saxon, Senior Research Fellow, Deakin University
Organization: Deakin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-399
Record Dates: First submitted 2021-06-21; First posted 2021-07-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Mental Health Wellness 1
Keywords: Prevention; Mental Health; Accountants; Small business owner
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Business advisor participants will be randomised to the treatment or control group using block randomisation. This process will be conducted by an external organisation who the participants are members of, so the trial investigators are blind to what study arm the participants are randomised to. The external organisation will provide potential participants with a computer generated unique ID, then order the IDs from highest to lowest, divide the list in half and allocate a block to the treatment or control arm. Allocation concealment will be achieved because the external organisation will not be able to predict the unique ID allocated to each participant before they are randomised to a group. The outcome assessor will be blinded to the participants study arm for the preliminary analysis. There are no subjective measures in this study. The participants will be blinded to their study group before they agree to participate to avoid self-selection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health First Aid and Relationship Building Training (MHFA+RBT) (Experimental): Mental Health First Aid training in conjunction with Relationship Building Training.
  Interventions: Behavioral: Mental Health First Aid and Relationship Building Training
- Mental Health First Aid (MHFA only) (Active Comparator): Mental Health First Aid training alone.
  Interventions: Behavioral: Mental Health First Aid

INTERVENTIONS:
Behavioral: Mental Health First Aid and Relationship Building Training — Relationship Building Training (RBT) is a 2 hour training session conducted live over zoom, that aims to equip business advisors the communications skills they need to enhance trustworthiness and quality of the relationship with their clients.
  Mental Health First Aid (MHFA) is a certified training program. It requires 5-7 hours of online course work followed by 2 x 2.5 hour live zoom sessions, that aims to enhance mental health literacy and teach the skills needed to identify the signs of mental health conditions and to have a conversation with a person who may need professional help.
  Two Booster sessions are delivered 1- and 3-months after the last MHFA session that aims to give participants the opportunity to consolidate their learning and share experiences applying the knowledge/skills gained.
  Participants will also invite 2-3 of their small-business entrepreneur (SME) clients to join the study and complete 3 surveys to provide feedback on the success of the program.
  Other Names: MHFA and RBT
  Arms: Mental Health First Aid and Relationship Building Training (MHFA+RBT)
Behavioral: Mental Health First Aid — Mental Health First Aid (MHFA) is a certified training program. It requires 5-7 hours of online course work followed by 2 x 2.5 hour live zoom sessions in addition to online reading, that aims to enhance mental health literacy and teach the skills needed to identify the signs of mental health conditions and to have a conversation with a person who may need professional help.
  MHFA online training is conducted two-weeks before the two MHFA sessions (with a 1 day break in between each MHFA). Two Booster sessions are delivered 1- and 3-months after the last MHFA session. The Booster sessions aims to give participants the opportunity to consolidate their learning and share experiences applying the knowledge/skills gained.
  Participants will also invite 2-3 of their small-business entrepreneur (SME) clients to join the study and complete 3 surveys to provide feedback on the success of the program.
  Other Names: MHFA alone
  Arms: Mental Health First Aid (MHFA only)

SUMMARY:
The financial state of a business and the mental health of the business owner are closely related. Thus, the devastating impact of COVID-19 on businesses means small-medium enterprises (SMEs) owners are particularly vulnerable to experiencing depression, anxiety and other mental health conditions (MHC). However, there is a tendency for SME owners to seek help about their financial concerns, rather than their mental wellbeing. For this reason, trusted business advisors (accountants, bookkeepers, coaches) who engage with their SME clients on a regular basis, are well-placed to provide advice about both the financial and mental health concerns of their SME clients.

To provide business advisors with the skills they need to have a conversation with their clients about their mental wellbeing and to encourage help-seeking where appropriate, mental health first aid (MHFA) training will be offered. And to help the business advisor forge a more trusting relationship with their client and provide higher quality advice that may alleviate their financial stresses, Relationship Building Training (RBT) will also be provided. Thus, the aim of this randomised control trial is to assess the additional benefit of combining RBT with MHFA compared with MHFA alone on the financial wellbeing of SME clients and the quality of their relationship with their business advisor.

DETAILED DESCRIPTION:
The widespread lockdown of broader society experienced around the world due to the COVID-190 pandemic is unprecedented. Businesses in a variety of sectors such as manufacturing, retail, and hospitality were closed due to lockdown rules, a decrease in demand, health concerns or other factors. Many of the closures are permanent because of the inability of business owners to pay ongoing expenses and market uncertainty.

Small to medium enterprises (SMEs) account for 99% of all businesses in Australia and at least 95% of enterprises in all OECD countries. SMEs provide an important contribution to Australia's growth in employment, with small businesses (including micro businesses) employing approximately 4.72 million people and accounting for 41 per cent of total employment. To help citizens survive the pandemic, the Australian government provided financial support to employees via Job Keeper and cash flow boosts to eligible businesses. Nevertheless, some SME owners reported losing up to 90% of their income and continue to face ongoing challenges, including market uncertainty, loss of international skilled workers, lending restrictions, extensive legislative reform. At the same time that they're dealing with an increasingly difficult external environment, SME owners also have to content with running a business including monitoring cash flow, managing staff, and ensuring the smooth administration of the business.

Of the challenges faced by SME owners, financial pressure represents a major source of psychological distress and is likely to explain why SME owners generally experience higher levels of stress and mental health disorders compared with the broader population. In Australia, 1 in 3 SMEs rated their mental health as poor to fair during the pandemic. Identifying the symptoms of depression early and encouraging help seeking are therefore critical and cost-effective methods for protecting and promoting wellbeing.

Mental health literacy programs have emerged as a key strategy for the early identification of diagnosable mental health problems. The strategy has proved to be popular in the frontline human service sectors (e.g., health care, social work) where MHFA can be used to help colleagues and members of the public who may be experiencing the signs of depression, anxiety and other mental health conditions (MHC's). However, little is known about the effectiveness of mental health literacy programs where SME owners are concerned. Reaching vast numbers of owner-managers in a systematic way is thought to be particularly difficult, partly because of the absence of viable intermediaries that have ongoing contact with this group, but also because of the typical characteristics of the SME owner's role (e.g., long working hours, burden of responsibility, isolation, obligation to work when sick), coupled with their lack of financial resources.

One sector that has the potential to act as an intermediary between small business and mental health services are business advisors, who include accountants, financial planners and financial counsellors. Business advisors are an important source of support for SME owners as their expertise is sought on a regular basis and clients can develop trusting, long-term relationships with their accountant. Previous work in this sector by Bond and colleagues has shown that MHFA training is an effective way of improving financial counsellors' ability to recognise mental health problems among clients and to provide appropriate support for help-seeking.

Despite the importance of mental health prevention programs like MHFA, these strategies are designed to reduce the impact of mental health conditions (i.e. secondary and tertiary prevention) rather than prevent them from occurring in the first instance (i.e., primary prevention). Longitudinal evidence causally implicates adverse psychosocial working conditions (e.g., excessive workloads, inadequate support) in the development of MHCs, such as depression. Thus, if business advisors can work to alleviate these stressors, they may also help prevent the onset of MHCs.

Therefore, the aim of the current project is to assess a new approach to undertaking MHFA training by incorporating a client-centred, Relationship Building Training (RBT) program that is designed to help business advisors better understand the business and personal needs of SME owners. If they better understand their needs, the business advisor can provide higher quality advice and in turn, reduce the financial stress of the SME owner. For any of this to happen, there needs to be a degree of trust generated between the business advisor and their SME client. According to Manister's trust equation, trustworthiness can be increased by improving how credible, reliable, and intimate you are and by decreasing your self-orientation. Thus, the RBT aims to equip the business advisor with the skills they need to enhance their intimacy and decrease their self-orientation. It is proposed, that if the business advisor builds a more trusting relationship with their clients that: i) it will reduce information asymmetry between the business advisor and client, enabling a better understanding of the SME's needs that leads to more personalised, tailed advice. In turn, this will alleviate the SME's financial stress and help prevent the onset of MHCs; and ii) it will allow the SME to feel more comfortable disclosing any financial concerns and/or mental health problems and when combined with the MHFA, the business advisor will better recognise the signs of MHCs and encourage them to seek help where appropriate.

Thus, this study represents a crucial next step in protecting the mental health of SME owners by assessing the incremental effectiveness of combining a primary prevention strategy (RBT) with the tertiary and secondary-level prevention approach of MHFA on the prevention of MHC's. It will be the first to assess the effectiveness of the approach through a randomised control trial (RCT) using a national sample of practising business advisors and their SME owner clients. Combined with the effectiveness trial, a process evaluation will be employed to identify the programs strengths and areas for improvement and to inform the expansion of this program to other sectors.

ELIGIBILITY:
Inclusion Criteria:

* Any qualified business advisor from Australia or New Zealand who provides business advice to a small-medium enterprise client (SME). Business advice refers to the information, guidance and/or assistance provided by an external adviser that either directly or indirectly helps to prevent/reduce the financial pressures experienced by SME owner-clients.
* The SME client must be the owner-manager/operator with 1-199 employees, including the owner-manager themselves.
* The business advisor must be in contact with their SME client at least 3 times a year.

Exclusion Criteria

* Any business advisor who has completed Mental Health First Aid within the last two years.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1599 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in the quality of the relationship between the small-medium business owner with the business advisor. | SMEs: Baseline, 5 + 11 months post training. BAs: Baseline, 1 + 5 months post training
  Quality of the Relationship Questionnaire aims to measure the SME owner's satisfaction with the level of attention they are receiving from the business advisor, and the business advisor's belief about how much attention they are providing. For the business advisors, 10 items will be used, four are from the Relationship Flourishing Scale (Fowers et al. 2016) that has a Cronbach's alpha of 0.93, and six are from a newly developed tool by principal investigators (AN, GT) with factor loadings of 0.81 to 0.87. The SME's will answer the latter six items. All items are on a 7-point Likert scale (1 strongly disagree, 7 strongly agree) with a higher total score indicating a stronger relationship.

SECONDARY OUTCOMES:
Process evaluation | Baseline, mid-training, 5-months post training
  The RE-AIM framework will be used to guide our evaluation of the intervention (Counting on U) (Glasgow 1999). RE-AIM stands for Reach, Effectiveness, Adoption, Implementation, and Maintenance. Field notes will be recorded, and structured interviews will be conducted with various stakeholders, including the business advisors, SME owners, trainers, and accounting/bookkeeper member bodies who will assist with the recruitment of business advisors. Process evaluation of Counting on U will help inform: 1) the future expansion and implementation of this program to various populations and 2) reveal both strengths and areas for improvement of the program strategies.
Change in psychological distress | SMEs: Baseline, 5 + 11 months post training. BAs: Baseline, 1 + 5 months post training
  Psychological Distress of the SME owners and business advisors will be measured using the Kessler 6 (K6) (Kessler et al 2002). This non-specific scale screens individuals for severe mental illness as defined as a K6 score ≥13. The K6 asks respondents, in the past four weeks how often did they feel the following: nervous, hopeless, restless or fidgety, worthless, depressed and felt that everything was an effort. For each question, a value of zero to four is assigned (0 none of the time, 4 all of the time), and a total score summed out of 24. The scale has demonstrated excellent internal consistency and reliability (Cronbach's alpha = 0.89) (Kessler et al 2002).
Change in MHFA knowledge | BAs: Baseline, 1 + 5 months post training
  Knowledge about mental health problems will be assessed using 18 questions adapted by Jorm et al (2010) that reviews information taught on day 1 and 2 of the Mental Health First Aid course. Questions consist of statements rated as Agree, Disagree or Unsure. The total score will be the number of questions answered correctly. An examples question is: "Half of all people who experience a mental illness have their first episode by age 18".
Change in confidence to provide MHFA | BAs: Baseline, 1 + 5 months post training
  Provision of Mental Health First Aid questions will include whether the business advisor had talked to a SME owner about their mental health problems over the past month using a 4-point Likert scale (1 never, 4 many times) (Jorm et al 2010). If they have talked with a SME owner client, they will be asked to indicate how many out of 12 actions they had taken. A score of 1 will be allocated to any action they have taken A Few or Many Times and summing these scores.
Change in stigmatisation | BAs: Baseline, 1 + 5 months post training
  Stigmatising attitude of the business advisors will be measured using six statements that queries their opinion of a person described in a vignette (personal stigma) (Reavley 2011). The modified vignette (Yap et al 2015) portrays a 35-year-old business owner who is showing signs of depression. An example of a personal stigma item is: "A problem like John's is a sign of personal weakness". Each item is scored on 5-point Likert scale (1 strongly agree, 5 strongly disagree) and the total score will be the number of items answered Agree or Strongly Agree.
Change in health seeking behaviour | SMEs: Baseline, 5 + 11 months post training. BAs: Baseline, 1 + 5 months post training
  Actual Health Seeking Behaviour questions will assess the SME owners and business advisor's behaviour of actively seeking assistance for mental health problems (Rickwood et al. 2005). The scale covers the informal, formal as well as physical and emotional aspect of help-seeking behaviour. The participant is asked to select from a list of people they have gone to for advice or help in the past two weeks.
Change in health, comfort, and happiness experienced by the individual (Quality of life). | SMEs: Baseline, 5 + 11 months post training. BAs: Baseline, 1 + 5 months post training
  Quality of Life questions will measure the general health of the business advisors and SME owners. The Short Form-12 questionnaire (SF-12) produces two summary scores - a mental component score (MCS-12) and a physical component score (PCS-12). This questionnaire has a test re-test reliability of 0.76 to 0.89 for the mental (MCS-12) and physical (PCS-12) health components (Ware 1996). Both components can discriminate among groups known to differ in their physical and mental conditions, yielding relative validities of 0.63 to 1.07 (Ware 1996). The answers are weighted, and the results are presented in reference to the United States population profile at the time of the original publication in 1994. A higher score for MCS and PCS indicates a better health state.
Change in financial wellbeing of small-medium enterprise (SME) owners | SMEs: Baseline, 5 and 11 month post-training.
  Financial Wellbeing Questionnaire (Prawitz 2006) consists of 8 items designed to gather information on how positively the SME owners view their financial situation. Each answer is scored from 1 to 10, and the total is summed and divided by 8. A higher score indicates no financial distress/ high financial well-being. The internal reliability of the scale is robust with a Cronbach's alpha of 0.956 indicating that the items contributing to the measurement of financial well-being, consistently yielded similar results. Factor loadings ranged from 0.83 to 0.93, indicating the measurement of only one latent construct.
Change in the degree of trust the small-medium business owner has in their business advisor | SMEs: Baseline, 5 + 11 months post training.
  Trust in Business Advisor Questionnaire measures the three elements of trust defined by Cherry et al. (2018): confidence, acting proactively and not exploiting vulnerabilities. In addition, the SME owner's confidence in the services (i.e., beyond compliance services) offered by the business advisor will be measured. Eleven questions will assess trust on a 5-point Likert scale (1 strongly disagree, 5 strongly agree) with a higher total score indicating a more trusting relationship. Factor loading for the items range from 0.43 to 0.95 and shows good reliability, with a Cronbach's alpha of 0.931 to 0.937.
Change in financial pressure | SMEs: Baseline, 5 + 11 months post training.
  Perceived Financial Wellbeing questions developed by Netemeyer et al 2018, asks the SME owners to consider how much they agree with 5 statements such as "I am behind with my finances". Their answers will be scored on a 5-point Likert scale (1 strongly agree, 5 strongly disagree) and a lower total mean score will indicate a more positive outlook. Perceived financial wellbeing is a strong predictor of overall well-being and has a Cronbach's alpha of 0.86 to 0.94 (Netemeyer et al. 2018).
Autonomy | BAs: Baseline + 5 months post training
  Autonomy will be measured using a 3-item scale that asks how much control the business advisor feels they have over their work and scored on a 5-point Likert scale (1 strongly disagree, 5 strongly agree) (Bakker et al, 2004, Karasek 1985). A mean score will be generated and a higher score indicating greater autonomy. The Cronbach's alpha is 0.68.
Emotional | BAs: Baseline, + 5 months post training
  Emotional Demands on the business advisors will be measured using the second version of the Copenhagen Psychosocial Questionnaire (Pejtersen et al, 2010). There are four items exploring how emotionally demanding they find their work, two items are measured on one 5-point Likert scale (1 never, hardly, 5 always) and two on a different 5-point Likert scale (1 to a very small extent, 5 to a large extent). The Cronbach's alpha is 0.87.
Workload | BAs: Baseline + 5 months post training
  Workload of the business advisors will be measuring using 3 items on a 5-point scale (1, not at all, 5 to a great extent) (Albrecht 2015, Karasek 1979). They will be asked their thoughts on statements such as "to what extent is there not enough time for you to do your job?" A mean score will be generated, and a higher score indicates a more demanding workload. The Cronbach's alpha is: 0.85 to 0.88.
Confidence and resilience | SMEs: Baseline, 5 + 11 months post training. BAs: 1 + 5 months post training
  Psychological Capital Short Form (PCQ-12) questionnaire measures wellbeing as a function of four emotions, two of which will be measured in the SME owners and business advisors: resilience and self-efficacy (Kamei et al 2018). Participants will respond to six statements on a 6-point Likert scale (1 strongly disagree, 6 strongly agree). PCQ-12 is designed for working adults and both resilience and self-efficacy statements are significantly correlated with measures of satisfaction with life, happiness and perceived stress (-0.36 to 0.50). The factor loadings of the questions range from 0.30 to 0.87.
Social support | SMEs: Baseline, 5 + 11 months post training. BAs: Baseline + 5 months post training
  Social Support questions assess the extent of emotional social support the participant receives from clients, family and friends, or colleagues and peers (Totterdal et al. 2006). The business advisors and SME owners will be asked two questions about each source: how easy is to talk to the people concerned and are the people concerned willing to listen to your problems. Responses are recorded on a 5-point Likert scale (1 not at all, 5 a great deal). The higher the score, the higher the social support. The Cronbach's alpha is 0.81.

CONTACTS AND LOCATIONS:
Overall Officials: Andew Noblet, PhD, Principal Investigator — Deakin University; George Tanewski, PhD, Principal Investigator — Deakin University
Locations (1):
- Deakin University, Burwood, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prawitz AD, Garman T, Sorhaindo B, O'Neill B, Kim J, Drentea P InCharge Financial Distress/Financial Well-Being Scale: Development, Administration, and Score Interpretation
- [Background] Mayer, R.C., Davis, J.H. and Schoorman, F.D. An integrative model of organizational trust. Academy of Management Review, 2005. 20(3): 709-734.
- [Background] Cherry M, McGrath D, Baumann C.Client intimacy & performance advice: Determinants of trust in the public accountant SME client relationship.Australasian Accounting, Business and Finance Journal. 2018; 12(1): 3-32
- [Background] Coulter K, Coulter R. Determinants of trust in a service provider: the moderating role of length of relationship. Journal of Services Marketing. 2002; 16(1): 35-50.
- [Background] Fowers BJ, Laurenceau JP, Penfield RD, Cohen LM, Lang SF, Owenz MB, Pasipandoya E. Enhancing relationship quality measurement: The development of the Relationship Flourishing Scale. J Fam Psychol. 2016 Dec;30(8):997-1007. doi: 10.1037/fam0000263. PMID 27918187
- [Background] Jorm AF, Kitchener BA, Fischer JA, Cvetkovski S. Mental health first aid training by e-learning: a randomized controlled trial. Aust N Z J Psychiatry. 2010 Dec;44(12):1072-81. doi: 10.3109/00048674.2010.516426. PMID 21070103
- [Background] Netemeyer RG, Warmath D, Fernandes D, Lynch GJ Jr. How Am I Doing? Perceived Financial Well-Being, Its Potential Antecedents, and Its Relation to Overall Well-Being Journal of Consumer Research. 2018; 45(1) 68-89,
- [Background] Totterdell P, Wood S, Wall T. An intra-individual test of the demands-control model: A weekly diary study of psychological strain in portfolio workers. Journal of Occupational and Organizational Psychology. 2006;79, 63-84
- [Background] Landells EM, Albrecht SL. Perceived Organizational Politics, Engagement, and Stress: The Mediating Influence of Meaningful Work. Front Psychol. 2019 Jul 10;10:1612. doi: 10.3389/fpsyg.2019.01612. eCollection 2019. PMID 31354596
- [Background] Albrecht SL. Job resources and employee engagement in a Chinese context: the mediating role of job meaningfulness, felt obligation and positive mood. International Journal of Business and Emerging Markets. January 2012
- [Background] Bakker AB, Demerouti E, Verbeke W. Using the job demands-resources model to predict burnout and performance. Human Resource Management. Spring 2004; 43(1):83-104
- [Background] Pejtersen JH, Kristensen TS, Borg V, Bjorner JB. The second version of the Copenhagen Psychosocial Questionnaire. Scand J Public Health. 2010 Feb;38(3 Suppl):8-24. doi: 10.1177/1403494809349858. PMID 21172767
- [Background] Albrecht SL. Challenge Demands, Hindrance Demands, and Psychological Need Satisfaction Their Influence on Employee Engagement and Emotional Exhaustion. Journal of Personnel Psychology 2015; 14(2):70-79
- [Background] Karasek RA. Job demands, job decision latitude, and mental strain: Implications for job redesign. Administrative Science Quarterly. 1979: 24: 285-308.
- [Background] Cocker F, Martin A, Scott J, Venn A, Sanderson K. Psychological distress, related work attendance, and productivity loss in small-to-medium enterprise owner/managers. Int J Environ Res Public Health. 2013 Oct 15;10(10):5062-82. doi: 10.3390/ijerph10105062. PMID 24132134
- [Background] Morgan AJ, Ross A, Reavley NJ. Systematic review and meta-analysis of Mental Health First Aid training: Effects on knowledge, stigma, and helping behaviour. PLoS One. 2018 May 31;13(5):e0197102. doi: 10.1371/journal.pone.0197102. eCollection 2018. PMID 29851974
- [Background] Martin A, Sanderson K, Scott J, Brough P. Promoting mental health in small-medium enterprises: an evaluation of the "Business in Mind" program. BMC Public Health. 2009 Jul 15;9:239. doi: 10.1186/1471-2458-9-239. PMID 19604351
- [Background] Bovopoulos N, LaMontagne AD, Martin A, Jorm A. Exploring the role of mental health first aid officers in workplaces: A qualitative study using case study methodology. Int J Workplace Health Manag. 2018;11(6):366-81
- [Background] Tetrick LE, Slack KJ, Da Silva N, Sinclair RR. A comparison of the stress-strain process for business owners and nonowners: differences in job demands, emotional exhaustion, satisfaction, and social support. J Occup Health Psychol. 2000 Oct;5(4):464-76. doi: 10.1037//1076-8998.5.4.464. PMID 11051529
- [Background] Bond KS, Chalmers KJ, Jorm AF, Kitchener BA, Reavley NJ. Assisting Australians with mental health problems and financial difficulties: a Delphi study to develop guidelines for financial counsellors, financial institution staff, mental health professionals and carers. BMC Health Serv Res. 2015 Jun 3;15:218. doi: 10.1186/s12913-015-0868-2. PMID 26037733
- [Background] LaMontagne AD, Martin A, Page KM, Reavley NJ, Noblet AJ, Milner AJ, Keegel T, Smith PM. Workplace mental health: developing an integrated intervention approach. BMC Psychiatry. 2014 May 9;14:131. doi: 10.1186/1471-244X-14-131. PMID 24884425
- [Background] LaMontagne AD, Milner AJ, Allisey AF, Page KM, Reavley NJ, Martin A, Tchernitskaia I, Noblet AJ, Purnell LJ, Witt K, Keegel TG, Smith PM. An integrated workplace mental health intervention in a policing context: Protocol for a cluster randomised control trial. BMC Psychiatry. 2016 Feb 27;16:49. doi: 10.1186/s12888-016-0741-9. PMID 26920745
- [Background] Noblet A, Lamontagne AD. The role of workplace health promotion in addressing job stress. Health Promot Int. 2006 Dec;21(4):346-53. doi: 10.1093/heapro/dal029. Epub 2006 Jul 31. PMID 16880197
- [Background] Tennant C. Work-related stress and depressive disorders. J Psychosom Res. 2001 Nov;51(5):697-704. doi: 10.1016/s0022-3999(01)00255-0. PMID 11728512
- [Background] Stansfeld S, Candy B. Psychosocial work environment and mental health--a meta-analytic review. Scand J Work Environ Health. 2006 Dec;32(6):443-62. doi: 10.5271/sjweh.1050. PMID 17173201
- [Background] IPA-Deakin SME Research Centre. Australian Small Business White Paper. Melbourne: 2018.
- [Background] Storey DJ. Understanding the small business sector: Routledge; 2016.
- [Background] Australian Bureau of Statistics (February 2021). 8165.0 Counts of Australian Businesses, including Entries and Exits. Commonwealth of Australia. https://www.abs.gov.au/statistics/industry/industry-overview/australian-industry/latest-release#data-download Accessed 20th February 2021.
- [Background] Ramsden M, Bennett R. The benefits of external support to SMEs: "Hard" versus "soft" outcomes and satisfaction levels. Journal of Small Business and Enterprise Development. 2005;12(2):227-43.
- [Background] icare and Everymind. White Paper: Can digital interventions help to improve mental health and reduce mental ill-health in small business? . NSW, Australia: 2017.
- [Background] Report Department for Industry, Science, Energy and Resources. "Small business and mental health: supporting small business when they are facing challenges". July 2020.
- [Background] Blackburn R, Carey P, Tanewski G. Business advice by accountants to SMEs: relationships and trust. Qualitative Research in Accounting & Management. 2018.
- [Background] Maister DH. The Trusted Advisor, Simon and Schuster, New York, 2001.
- [Background] Yap MB, Reavley NJ, Jorm AF. Is the use of accurate psychiatric labels associated with intentions and beliefs about responses to mental illness in a friend? Findings from two national surveys of Australian youth. Epidemiol Psychiatr Sci. 2015 Feb;24(1):54-68. doi: 10.1017/S2045796013000607. Epub 2013 Nov 7. PMID 24229559
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Reavley NJ, Jorm AF. Stigmatizing attitudes towards people with mental disorders: findings from an Australian National Survey of Mental Health Literacy and Stigma. Aust N Z J Psychiatry. 2011 Dec;45(12):1086-93. doi: 10.3109/00048674.2011.621061. Epub 2011 Oct 24. PMID 22023236
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Kamei H, Ferreira MC, Valentini F, Peres MFP, Kamei PT, Damásio BF. Psychological Capital Questionnaire - Short Version (PCQ-12): evidence of Validity of The Brazilian Psico-USF, Bragança Paulista. 2018 23(2): 203-214
- [Background] Karasek R. Job content instrument: Questionnaire and user's guide, revision 1.1. Los Angeles: University of Southern California. 1985
- [Background] Karasek RA. Job demands, job decision latitude and mental strain: Implications for job redesign. Administrative Science Quarterly. 1979; 24, 285-308.
- [Background] Albrecht SL, Su MJ. Job resources and employee engagement in a Chinese context: the mediating role of job meaningfulness, felt obligation and positive mood. Int. J. Business and Emerging Market. 2012; 4(4).
- [Background] Noblet AJ, LaMontagne AD. The challenges of planning, implementing and evaluating interventions. In: Cartwright S, Cooper CL, editors. The Oxford Handbook of Organizational Well-Being. Oxford: Oxford University Press; 2009: 466-96.
- [Derived] Saxon L, Bromfield S, Leow-Taylor SH, Vega CE, Berk M, LaMontagne AD, Martin AJ, Mohebbi M, Nielsen K, Reavley NJ, Walker A, Conway A, de Silva A, Memish K, Rossetto A, Tanewski G, Noblet A. Counting on U training to enhance trusting relationships and mental health literacy among business advisors: protocol for a randomised controlled trial. BMC Psychiatry. 2022 Jun 15;22(1):400. doi: 10.1186/s12888-022-04034-7. PMID 35705927